CLINICAL TRIAL: NCT02420548
Title: Preventing Drug Use and Risk Behaviors in Adolescent Girls
Brief Title: Safe, Healthy, Adolescent Relationships and Peers
Acronym: SHARP-Teen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Oregon Social Learning Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10312013.040; 1P50DA035763 (NIH)
Record Dates: First submitted 2015-04-14; First posted 2015-04-20 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Juvenile Delinquency Unspecified; Risk Behavior; Adolescent Behavior; Sexual Behavior; Drug Use
MeSH Terms: conditions — Risk-Taking; Adolescent Behavior; Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as Usual (Active Comparator): Participants continue with any services they may be receiving outside of the study.
  Interventions: Behavioral: Services as Usual
- Parent Ed. and Youth Skills Coaching (Experimental): The experimental intervention will have two components: (1) a caregiver parenting group, including all caregiver types (biological, foster, kinship), that meets weekly for 90-minutes for four months, focused on increasing parenting skills, and (2) a Life Coach component where trained and supported skills coaches meet individually with youth weekly for 60 minutes over the same four-month period to build the girls' social skills and peer/partner relationships skills.
  Interventions: Behavioral: Parent Ed. and Youth Skills Coaching; Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: Parent Ed. and Youth Skills Coaching — The experimental intervention will have two components: (1) a caregiver parenting group, including all caregiver types (biological, foster, kinship), that meets weekly for 90-minutes for four months, focused on increasing parenting skills, and (2) a Life Coach component where trained and supported skills coaches meet individually with youth weekly for 60 minutes over the same four-month period to build the girls' social skills and peer/partner relationships skills.
  Arms: Parent Ed. and Youth Skills Coaching
Behavioral: Services as Usual — Services as usual as provided by community service organizations from which the sample was drawn.

SUMMARY:
The Safe, Healthy, Adolescent Relationships and Peers study seeks to understand some of the factors that contribute to the behaviors and health of teen girls, such as girl's friendships, their dating behaviors, their risk-taking behaviors, and their knowledge about how to make healthy choices. This study will inform us on ways to help teen girls engage in safe and healthy relationships and adjustment.

DETAILED DESCRIPTION:
Initiation of drug use and participation in sexual-risk behaviors such as having multiple sexual partners, unprotected sexual intercourse, and intercourse with drug users are all too common among girls with at-risk histories, such as those who have experienced poverty, abuse, neglect, or been in the juvenile justice system. Studies consistently find that these girls have disproportionately high rates of these problems that, in addition to increasing risk for negative outcomes, have other costly sequelae such as drug addiction, early pregnancy, sexually-transmitted infections (STIs) and HIV contraction, delinquency, and early mortality (e.g., Santelli et al., 2001; Stueve et al., 2005). In our prior work, the investigators showed that the investigators could prevent early onset sexual intercourse and tobacco and marijuana initiation in pre-teen girls in foster care. Although this intervention, delivered to girls who were 11-years old and had not yet entered middle school, demonstrated efficacy, the investigators know very little about how to prevent the more serious and costly sexual-risk and illicit drug use behaviors in at-risk girls during the high school years, a period of risk for engagement in such behaviors. This study builds from this prior work to develop a new intervention for teenage girls with early adversity.

ELIGIBILITY:
Inclusion Criteria:

* reside in Lane County and within 70 miles of the University of Oregon
* have a current caregiver
* both girl and caregiver are fluent in English

Exclusion Criteria:

* are medically fragile
* have a significant developmental disability
* have graduated from high school or have a General Educational Diploma (GED)

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Delinquency measured by official arrest records and standardized questionnaires | Up to 12 months
  Reduction in delinquent behaviors for teens participating in the intervention arm measured by official arrest records and standardized questionnaires, including the Youth Symptom inventory, the Elliott Self-report Delinquency Scale, the Achenbach System of Empirically Based Assessment, and the Parent Daily Report.
Sexual Risk Behavior | Up to 12 months
  Reduction in high risk sexual behaviors for teens participating in the intervention arm measured by standardized questionnaires, including Partner and Peer Behavior, Conflict in Adolescent Dating, Sexual Health Scale, and the Parent Daily Report.

SECONDARY OUTCOMES:
Parenting measured by change in parenting practices for parents participating in the intervention arm measured by standardized questionnaires | Up to 12 months
  including the Monitoring and Parent-Child Relationship, the Parent Practices Scale, the Parent Daily Report, and the Unrevealed Differences Questionnaire.
Substance Use | Up to 12 months
  Reduction in substance use for teens participating in the intervention arm measured by urine analysis and standardized questionnaires, including the Youth Symptom Inventory, the World Health Organization Composite International Diagnostic Interview, and the Parent Daily Report.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Leve, PhD, Principal Investigator — University of Oregon; Patti Chamberlain, PhD, Principal Investigator — Oregon Social Learning Center; Rohanna Buchanan, PhD, Study Director — Oregon Social Learning Center
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Completely de-identified data shared. Interested investigators must secure IRB approval or waiver from their institution and cerfiy that they will not attempt to discern the identity of any participant.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: December 2021. No specific end date
Access Criteria: Email: leve@uoregon.edu

REFERENCES:
- [Result] Horn SR, Leve LD, Levitt P, Fisher PA. Childhood adversity, mental health, and oxidative stress: A pilot study. PLoS One. 2019 Apr 26;14(4):e0215085. doi: 10.1371/journal.pone.0215085. eCollection 2019. PMID 31026258
- [Result] Clark M, Buchanan R, Kovensky R, Leve LD. Partner influences on young women's risky drug and sexual behavior. Reprod Health. 2018 Sep 15;15(1):156. doi: 10.1186/s12978-018-0598-0. PMID 30219076
- [Result] Clark M, Buchanan R, Leve LD. Young Women's Perspectives of Their Adolescent Treatment Programs: A Qualitative Study. Int J Environ Res Public Health. 2018 Feb 22;15(2):373. doi: 10.3390/ijerph15020373. PMID 29470424
- [Result] Kovensky R, Anderson D, Leve LD. Early Adversity and Sexual Risk in Adolescence: Externalizing Behaviors as a Mediator. J Child Adolesc Trauma. 2019 Aug 7;13(2):173-184. doi: 10.1007/s40653-019-00278-w. eCollection 2020 Jun. PMID 32549929

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02420548/Prot_SAP_000.pdf